# Effect of in vitro fertilisation (IVF) hormonal therapy on metabolic, endocrine and inflammatory status in IVF-conceived pregnancy

NCT03426228

#### Chapter 1: Aim of the study and Objectives

- 1. To explore the short-term effects of IVF hormonal therapy on maternal metabolic and inflammatory status, including:
  - i. Risk of glucose intolerance and insulin resistance
  - ii. Risk of other metabolic, endocrine and inflammatory disturbances (including lipid profile, gut microflora and thyroid function)
- 2. To identify possible early predictors of GDM and other metabolic-related adverse outcomes in IVF-conceived pregnancies.

#### Chapter 2: General Methods

#### 2.1. Ethics and Consents

Approval to conduct the study was first granted by the University of Warwick's Biomedical and Scientific Research Ethics Sub-Committee (BSREC). The study protocol was also reviewed by the two main health authorities in the UAE.

#### 2.2. Study Design

The presented study is a longitudinal quantitative cohort study (non-experimental), whereby blood samples were collected at different stages during IVF therapy.

#### 2.3. Study Setting

The study took place at in three fertility clinics in the UAE. At the clinics, pre- and post-fertility treatments and in-house obstetric facilities are provided, including blood tests, scans, IVF procedures and in-house genetic testing. Most patients are followed up to the point of delivery.

#### 2.4. Study Population

- ➤ **Pregnant group**: received IVF therapy and tested <u>positive</u> for pregnancy at 4 weeks, and continued taking IVF hormonal therapy until 12 weeks of pregnancy.
- ➤ *Non-pregnant*: received IVF therapy and tested <u>negative</u> for pregnancy at 4 weeks, and stopped taking IVF hormonal therapy at that point.

#### 2.5. Sampling Technique

The non-probability convenience sampling method was used to recruit participants for the study. Patients who were to start a fresh IVF treatment at any of the IVF Clinic branches and meeting the inclusion criteria were eligible to participate.

#### 2.6. Study Protocol

After an overnight fast of 8 hours, there was collection of 10 ml of blood at four pre-defined time points during the IVF protocol:

- 1. **Phase 1** At baseline, egg maturation (starting IVF therapy)
- 2. *Phase 2* Week 2 Egg retrieval (OPU procedure)
- 3. *Phase 3* Week 4 At pregnancy test (β-HCG test)
- 4. **Phase 4** Week 12 (one week after completing IVF hormonal therapy for pregnant group).

#### 2.7. Blood Tests

A trained nurse was in charge of measuring anthropometrics and clinical parameters (e.g. weight and blood pressure), in addition to taking fasting blood samples. The socio-demographics, medical and pregnancy histories of each patient

were recorded in their file. Blood tests were conducted at in the phlebotomy room and transferred to the lab (in-house) for analysis. Tests results were available on the clinics internal server at the end of each day.

Table 1: List of Blood Tests at Each Stage of the Study

| Type of Tests | Phase 1-<br>Baseline<br>(Start IVF<br>treatment) | Phase 2-<br>Week 2 (Egg<br>retrieval) | Phase 3-<br>Week 4 (β-<br>HCG test) | Phase 4-<br>Week 12<br>(Final) |
|---|---|---|---|---|
| Female reproductive<br>hormones: FSH, LH,<br>oestrogen,<br>progesterone | ٧ | V | ٧ | |
| HbA1c | ٧ | | | ٧ |
| Fasting glucose | ٧ | ٧ | ٧ | ٧ |
| Fasting insulin | ٧ | ٧ | ٧ | ٧ |
| TSH | ٧ | | | ٧ |
| Fasting lipid profile | ٧ | | | ٧ |
| Adiponectin | ٧ | | | ٧ |
| LBP | ٧ | | | ٧ |
| β-HCG pregnancy | ٧ | | ٧ | |
| Body weight | ٧ | | | ٧ |

<sup>\*</sup>Green highlight represents stage where non-pregnant vs. pregnant women groups were distinguished; FSH: follicle-stimulating hormones; LH: luteinizing hormone; HbA1c: glycated haemoglobin A1c; TSH: thyroid-stimulating hormone; LBP: lipopolysaccharide binding protein;  $\beta$ -HCG: beta-human chorionic gonadotrophin

### Appendix 1. Anthropometrics and Medical History Questionnaire

Effects of fertility drugs on glucose homeostasis, and other metabolic parameters on patients undergoing In Vitro Fertilisation (IVF) NCT03426228

| Subject Name:<br>Telephone No:<br>E-mail: | | |
|-------------------------------------------|-----------|-----------|
| Age | | |
| Height | | |
| Weight | | |
| BMI | | |
| Nationality | | |
| Smoking | | |
| Parity | | |
| Past Illness and | Surgeries | |
| Drug History | | |
| Family History | | |
| Women Health | | |
| Cycle: | Regular | Irregular |

| History of GDM: |
|-----------------------------|
| <b>Previous IVF trials:</b> |

**Blood Analysis** 

| Diodu Alialysis | | |
|-------------------------|-------------|-----------|
| Туре | Level/ Unit | Frequency |
| Fasting glucose | | 4 times |
| Serum insulin | | 4 times |
| Lipid profile | | Twice |
| FSH, LH | | 4 times |
| Oestrogen, Progesterone | | 4 times |
| Beta-HCG | | Once |

#### Appendix 2. Participants Study Tests

## Effects of fertility drugs on glucose homeostasis, and other metabolic parameters on patients undergoing In Vitro Fertilisation (IVF) NCT03426228

#### IVF MEDICATION & METABOLIC PARAMETERS

| Baseline | Week2 | Week 2 | Week 4 | Week 12 |
|---|---|---|---|---|
| Start IVF Therapy | Pre-OPU | Embryo Transfer | +/- β-HCG | Final |
| A1C Fasting glucose Serum insulin Lipid profile Hormonal Profile (AMH, LH, FSH, progesterone, oestrogen) TSH LBP Adiponectin | Fasting glucose<br>Serum insulin<br>Hormonal profile (LH,<br>progesterone,<br>oestrogen) | Hormonal Profile<br>(progesterone,<br>oetrogen) | Fasting glucose<br>Serum insulin<br>Hormonal profile<br>(progesterone,<br>oestrogen, β-HCG) | HbA1c Fasting glucose Serum insulin Lipid profile TSH LBP Adiponectin |